CLINICAL TRIAL: NCT06613178
Title: Intravenous Acetaminophen After Cardiac Surgery
Brief Title: Intravenous Acetaminophen After Cardiac Surgery - Definitive Study
Acronym: IVACS
Status: Recruiting | Phase: Phase 4 | Type: Interventional
Sponsor: McGill University Health Centre/Research Institute of the McGill University Health Centre (Other)
Collaborators: Laval University (Other); University of British Columbia (Other); St. Boniface Hospital (Other); University of Ottawa (Other); Trillium Health Centre (Other); Université de Montréal (Other); Sunnybrook Health Sciences Centre (Other)
Responsible Party: Principal Investigator, magder sheldon, Principle Investigator, McGill University Health Centre/Research Institute of the McGill University Health Centre
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Prevention
Other Study IDs: MUHC-ACETAMINOPHEN FULL STUDY
Record Dates: First submitted 2024-03-01; First posted 2024-09-25 (Actual); Last update posted 2024-09-25 (Actual); Status verified 2024-07

CONDITIONS: Post Operative Delirium; Post Operative Pain; Post-Op Complication; Post-cardiac Surgery
Keywords: pain; post-operative care; cardiac surgery; narcotic; acetaminophen
MeSH Terms: conditions — Emergence Delirium; Pain, Postoperative; Postoperative Complications; Pain | interventions — Acetaminophen

STUDY DESIGN:
Intervention Model Description: randomized double blind double dummy two arm study
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Masking Description: Quadruple. blinded medication with codes kept by pharmacy director
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- Oral Placebo (Active Comparator): Subject receives active intravenous acetaminophen and oral placebo acetaminophen
  Interventions: Drug: acetaminophen
- Oral Acetaminophen (Placebo Comparator): Subject receives placebo IV fluid (saline) and active oral acetaminophen
  Interventions: Drug: acetaminophen

INTERVENTIONS:
Drug: acetaminophen — Patient receive IV acetaminophen (and oral placebo) or placebo IV acetaminophen and oral acetaminophen. All drugs are blinded
  Other Names: placebo

SUMMARY:
Double blind, double dummy trial of the use of IV acetaminophen versus oral acetaminophen for the prevention of delirium after cardiac surgery. The underlying hypothesis is that better pain control and less use of narcotics will lead to a lower incidence of delirium from day 1 to 7 following cardiac surgery. Other important secondary outcomes are the total use of narcotics, ICU and hospital stay, improved cognitive function at 6 months and 1 year post surgery, NSAID use at each centre and associated NSAID complications.

DETAILED DESCRIPTION:
Patients > or equal to 18 years of going for elective cardiac surgery will be randomized to receive IV either IV acetaminophen and an oral placebo acetaminophen or an IV placebo acetaminophen (saline) and oral acetaminophen every 6 hours for 48 hours after cardiac surgery. the study will be performed at 8 large Canadian cardiac surgery centres. All other therapy will be as per standard procedures (pragmatic) at the institutions including including use of their standard opioid protocol. The primary end-point is the development of delirium as assessed by Confusion Assessment Method in the Intensive Care unit (CAMICU) and the CAM on the regular floor unit for up to 7 days after surgery or discharge if it is sooner. Other measures are change from pre-operative cognitive function as assessed by the Montreal Cognitive Assessment score (MoCA) at 6 months and 1 year, numeric pain score, total opioid use, hospital and ICU length of stay. Use of opioids and pain score at 1 year also will be assessed. Patients will be stratified by site and sex.

We also will assess use of NSAID, specifically ketorolac, and any NSAID associated events.

ELIGIBILITY:
Inclusion Criteria:

greater or equal to 18

* elective cardiac surgery
* stable pre-operative
* aorto-coronary bypass with or without 1 valve replacement.

Exclusion Criteria:

Refusal by surgeon Requested late extubation by surgeon or anesthesia Intra-aortic balloon pump Mechanical cardiac support Sensitivity to acetaminophen Psychiatric history with current active treatment Alzheimer's disease Seizure in previous 6 months Recent history of alcohol misuse Cognitive impairment

-

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 1100 (Estimated)
Dates: Start 2024-07-02 (Actual); Primary Completion 2027-07-01 (Estimated); Study Completion 2027-12-15 (Estimated)

PRIMARY OUTCOMES:
post operative delirium | up to 7 days
  measured with CAMICU or CAM

SECONDARY OUTCOMES:
total use of opioids | up to 7 days
  measured for 7 days or until hospital discharge
Cognitive function at 6 months and 1 year | 6 months and 1 year
  Measured with Montreal Cognitive assessment score.
Time in intensive care unit | up to 7 days
  measured in hours
time in hospital | up to 7 days
  measured in days
time to extubation | up to 7 days
  measured in hours

CONTACTS AND LOCATIONS:
Locations (8):
- Canada (8):
  - University of British Columbia, Vancouver, British Columbia
  - University of Manitoba, Winnipeg, Manitoba
  - Trillium Health Centre, Mississagua, Ontario
  - University of Ottawa, Ottawa, Ontario
  - Sunnybroook Health Centre, Toronto, Ontario
  - McGill Universtiy Health Centre, Montreal, Quebec
  - Universite Montreal, Montreal, Quebec
  - University of Laval, Québec, Quebec

IPD SHARING:
Plan to Share IPD: No
If the investigators of PANDORA complete their study we would request to combine our studies in a meta-analysis